CLINICAL TRIAL: NCT04873986
Title: A New Clinical Tool for Scoliosis Risk Analysis: Scoliosis Tele-Screening Test
Brief Title: Scoliosis Tele-Screening Test
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, FİLİZ TUNA, Assoc Prof, Trakya University
Other Study IDs: TÜTF-BAEK 2020/287
Record Dates: First submitted 2021-05-02; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Scoliosis; Posture Disorders in Children
Keywords: Scoliosis screening; Tele-medicine; virtual assessment; posture
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Scoliosis Tele-Screening Test — Scoliosis Tele-Screening test will be applied to children by parents at home. Participants with moderate and high risks will be invited to the physical examination to the centers or virtual assessment via e-mail. The researchers will be evaluated the TRACE and Adams' test from the photo and sent their opinions to the parents via e-mail.

SUMMARY:
A new Scoliosis Tele-Screening Test (STS-Test) was developed by a study group of the "Scoliosis Research and Treatment Association Turkey". It will be sent to the families of schoolchildren by e-mail in Turkey. Participants with moderate and high risk for scoliosis according to the result of this test will be invited to the physical examination by the scoliosis specialists, if it is not possible, they will be evaluated via tele-medicine. Participants with moderate and high risks will be invited to the physical examination to the centers designated as research centers. Families who could not reach these centers will be asked to take pictures of their children according to the given instruction. They will be asked to send this photo to the researchers by e-mail. The researchers will be evaluated the TRACE and Adams' test from the photo and sent their opinions to the parents via e-mail. If this virtual analysis made by the expert suggests a suspicion of scoliosis, it will be recommended to see a specialist as soon as possible.

The aim of this study is to evaluate the validity and reliability of this novel scoliosis tele-screening test. A secondary aim is to investigate the coherence of this new test between scoliosis physician and parent when applied to the same child. Specificity, sensitivity, negative predictive value, positive predictive value, and test accuracy will be calculated for the Scoliosis Tele-Screening Test. Correlation between STS-Test and Trace, Adams' test, and physician diagnosis will be analyzed.

DETAILED DESCRIPTION:
Scoliosis is a three-dimensional spinal and trunk deformity. Adolescent Idiopathic Scoliosis prevalence is 3,1% in females and 1,5% in males in Turkey. Most of the cases are asymptomatic, therefore screening programs are very crucial for early diagnosis especially for cases in risky ages. Early diagnosis provides the early treatment.

Aesthetic evaluation of the trunk is one of the important components of Idiopathic Scoliosis and aesthetic appearance which is the main complaint of the patients and family is the primary aim of the conservative and operative treatment. There are some tools that evaluates postural asymmetries like Trunk Aesthetic Clinical Evaluation which evaluates the shoulder, scapula, waist, and hemithorax and known as a reliable instrument for everyday clinical evaluation and to monitor aesthetic changes achieved with treatment.

A scoliosis screening test has been developed in which families with restricted access to the hospital and healthcare professionals due to the Covid-19 pandemic, can evaluate their children in terms of scoliosis risk without applying to any health institution. A study group of subject experts was formed within the "Scoliosis Research and Treatment Association Turkey". This new tele-screening test could be easily applied by parents at a home in different times, give information about the results to the implementer just after the evaluation. Researchers discussed how to evaluate the spine for scoliosis in a virtual environment and were created a visual screening test. In the scoring of the STS-Test, the images related to the body asymmetry of patients with scoliosis with different deformities characteristics in the common database of these experts were analyzed and scoring was created by expert opinion and consensus.

Scoliosis risk was determined by considering the visual body asymmetries in the shoulder, thorax, waist, and pelvis, in addition, Adams' test. For the girls, female gender and time since menarche as a risk factor were included in the total score. In STS-Test scoring, the positive Adams' test is 4 points for both genders; the presence of family history related to scoliosis is 1 point; female gender was as 1 point; no menarche, or time less than 1-year since menarche for girls, was determined as 1 point. In the scoring of the other items, the anterior shoulder levels and height difference in the pelvis were scored as 2 points; if there was asymmetry in the images of the items including shoulder level difference from the posterior, scapula asymmetry, pelvic shifting to one side and height difference in the pelvis, they were scored as 1 point, and if symmetrical or not able to make a decision, it was scored as 0 points. Scoliosis Tele-Screening Test consists of a total of 23 Likert-type questions; 5 questions about the sociodemographic characteristics of the parents, 3 questions on the knowledge/awareness level regarding scoliosis, 3 questions on the risk factors related to scoliosis development, 7 questions about the cosmetic deformities that scoliosis may cause/can reveal, and 5 questions the satisfaction of the parent/evaluator. The total score for risk groups is based on 7 questions about the cosmetic deformities caused by scoliosis and 3 questions regarding the risk factors associated with scoliosis development. The total score is obtained by summing up the scores from 10 questions of these two sections. The total score is categorized as low, medium, and high risk, and the risk groups differ for males and females. 0-4 points are low, 5-11 points are medium, and 12-15 points are considered a high-risk group for girls in the total score. 0-3 points are low, 4-8 points are medium, and 9-13 points are considered high risk group for males in the total score.

The final version of the test was shared on the website of the Scoliosis Research and Treatment Association Turkey and social networks. After the parent/evaluator completed the test, an e-mail containing information about the test, scoliosis risk score, and recommendations was sent with an automatic reply. Participants with moderate and high risks will be invited to the physical examination to the centers designated as research centers. Families who could not reach these centers will be asked to take pictures of their children according to the given instruction. They will be asked to send this photo to the researchers by e-mail. The researchers will be evaluated the TRACE and Adams' test from the photo and sent their opinions to the parents via e-mail. If this virtual analysis made by the expert suggests a suspicion of scoliosis, it will be recommended to see a specialist as soon as possible. The patients who could apply to the center will be examined by the physician, evaluated cosmetically according to TRACE, and Adams' test will be performed. Suspicion of scoliosis will be confirmed by spine radiography. Patients with a Cobb angle ≥10° in any segment of the spine will be considered to have scoliosis. The location, direction, and angle of scoliosis will be recorded from the spine radiographs.

ELIGIBILITY:
Inclusion Criteria:

* healthy children who agree to voluntarily participate in the study by parents and theirself
* parents must be literate and have the ability to use the internet

Exclusion Criteria:

* neurological disease
* spine surgery history
* any disease that prevents standing position
* any cognitive impairment or communication problem

Ages: 9 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Schoolchildren age between 9-16 in Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 865 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Scoliosis Tele-Screening Test | through study completion, an average of 1 year
  Test Accuracy will be obtained using the formula below Test Accuracy/Power = ((TP+TN) / (TP+TN+FP+FN)) * 100 (TP: True positive, TN: True negative, FN:False negative, FP: False positive) Referral criteria for the accuracy of STS-Test based on Adams' test additionally clinician examination
To investigate the consistency between researchers' assessment and the results of the Scoliosis Tele-Screening Test by the parents for the same case | through study completion, an average of 1 year
  The agreement between the risk analyzes obtained with the STS-Test performed by the parents and the face-to-face spine assessment by a doctor will be determined. Pearson correlation coefficient will be used to investigate the correlations between parents(via the STS-Test score) and physician assessment. Correlation between parameters will be interpreted as follows: r=0-0.19 a very weak correlation, r=0.20-0.39 weak correlation, r=0.40-0.59 moderate correlation, r=0.60-0.79 strong correlation and r=0.80-1 very strong correlation.

SECONDARY OUTCOMES:
Trunk Aesthetic Clinical Evaluation score | Baseline
  Trunk Aesthetic Clinical Evaluation (TRACE) is a clinical tool developed for the evaluation of trunk asymmetries of patients with scoliosis by physicians or therapists. TRACE is a scale that evaluates asymmetry in shoulders, scapula, waist and hemithorax in 4 items and gives a global score that can reflect the clinical change over time. It is scored between 0-2 points for shoulder asymmetry, hemithorax asymmetry, scapula asymmetry, and 0-4 points for waist asymmetry. The total score is obtained by adding 1 point to the total scores of the 4 items, and scoring varies between 1 and 12 points. High scores are associated with increased body asymmetry.
Adams' Forward Bending Test | Baseline
  Adams' Forward Bending Test (FBT) is a clinical test that is frequently performed to reveal the suspicion of scoliosis in scoliosis screening. FBT shows the rib hump deformity caused by the vertebrae and ribs affected by scoliosis when the patient is in the forward bending position. It will recorded as positive or negative

CONTACTS AND LOCATIONS:
Overall Officials: Hurriyet Yilmaz, Prof, Study Director — Haliç University; FİLİZ TUNA, Assoc Prof, Principal Investigator — Trakya University; Aslıhan Kuşvuran Özkan, MD, Principal Investigator — Özel Özülkü Medical Center; Sibel Özdoğan, MD, Principal Investigator — Yıldız Medstar Hospital; Zeynep Turan, MD, Principal Investigator — Koç University; Ahsen Büyükaslan, PT, MSc, Principal Investigator — Formed Scoliosis Brace and Treatment Center; Hande Tunç, PT, MSc, Principal Investigator — Formed Scoliosis Brace and Treatment Center
Locations (1):
- Halic University, Istanbul, Beyoğlu/İstanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It was not planned to share individual participant data

REFERENCES:
- [Background] Prowse A, Pope R, Gerdhem P, Abbott A. Reliability and validity of inexpensive and easily administered anthropometric clinical evaluation methods of postural asymmetry measurement in adolescent idiopathic scoliosis: a systematic review. Eur Spine J. 2016 Feb;25(2):450-66. doi: 10.1007/s00586-015-3961-7. Epub 2015 Apr 28. PMID 25917824
- [Background] Zaina F, Negrini S, Atanasio S. TRACE (Trunk Aesthetic Clinical Evaluation), a routine clinical tool to evaluate aesthetics in scoliosis patients: development from the Aesthetic Index (AI) and repeatability. Scoliosis. 2009 Jan 20;4:3. doi: 10.1186/1748-7161-4-3. PMID 19154604
- [Background] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499
- [Background] Yilmaz H, Zateri C, Kusvuran Ozkan A, Kayalar G, Berk H. Prevalence of adolescent idiopathic scoliosis in Turkey: an epidemiological study. Spine J. 2020 Jun;20(6):947-955. doi: 10.1016/j.spinee.2020.01.008. Epub 2020 Jan 20. PMID 31972303
- [Background] Negrini S, Grivas TB, Kotwicki T, Maruyama T, Rigo M, Weiss HR; Members of the Scientific society On Scoliosis Orthopaedic and Rehabilitation Treatment (SOSORT). Why do we treat adolescent idiopathic scoliosis? What we want to obtain and to avoid for our patients. SOSORT 2005 Consensus paper. Scoliosis. 2006 Apr 10;1:4. doi: 10.1186/1748-7161-1-4. PMID 16759352
- [Background] Donaldson S, Stephens D, Howard A, Alman B, Narayanan U, Wright JG. Surgical decision making in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2007 Jun 15;32(14):1526-32. doi: 10.1097/BRS.0b013e318067dc75. PMID 17572623
- [Background] Negrini S, Donzelli S, Di Felice F, Zaina F, Caronni A. Construct validity of the Trunk Aesthetic Clinical Evaluation (TRACE) in young people with idiopathic scoliosis. Ann Phys Rehabil Med. 2020 May;63(3):216-221. doi: 10.1016/j.rehab.2019.10.008. Epub 2019 Dec 6. PMID 31816447